CLINICAL TRIAL: NCT05302258
Title: Noninvasive Assessment of Hepatic Steatosis by Using Attenuation Imaging in Children
Brief Title: Attenuation Imaging in Hepatic Steatosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ATI
Record Dates: First submitted 2022-03-18; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hepatic Steatosis; Obesity, Childhood; Ultrasonography
MeSH Terms: conditions — Fatty Liver; Pediatric Obesity | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obesity: BMI of 95 th percentile or more
  Interventions: Diagnostic Test: Attenuation imaging in ultrasonography
- Normal weight: BMI of 85 th percentile or less
  Interventions: Diagnostic Test: Attenuation imaging in ultrasonography

INTERVENTIONS:
Diagnostic Test: Attenuation imaging in ultrasonography — Attenuation imaging in ultrasonography

SUMMARY:
For obese and normal-weight children, the investigators assess the diagnostic performance of attenuation imaging (ATI) in the detection of hepatic steatosis in children.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 85th percentile or less

Exclusion Criteria:

* congenital anomaly including heart, intestine, kidney
* acute hepatitis
* congenital hepatic anomaly

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Obese and normal-weight children
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-04-14 (Estimated); Primary Completion 2022-12-14 (Estimated); Study Completion 2022-12-14 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of attenuation imaging | through study completion, an average of 1 year
  The diagnostic performance of attenuation imaging in US in the detection of hepatic steatosis